CLINICAL TRIAL: NCT03861585
Title: Attentional and Emotional Processing of Complex Visual Scenes in Children With Attention Deficit Disorder With or Without Hyperactivity
Brief Title: Emotional Information Processing in Attention Deficit Disorder With or Without Hyperactivity
Acronym: TIVE-TDA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Lenval (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 18-HPNCL-07
Record Dates: First submitted 2019-02-21; First posted 2019-03-04 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2019-05

CONDITIONS: Attention Deficit Disorder With Hyperactivity; Attention Deficit Disorder Without Hyperactivity
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- semantic group (Experimental): Half of the participants (named the "semantic group") perform a semantic categorisation task.
  Interventions: Other: Semantic group
- emotional group (Experimental): Half of the participants (named the "emotional group") perform an emotional evaluation task.
  Interventions: Other: Emotional group

INTERVENTIONS:
Other: Semantic group — The "semantic task" has to categorise semantically (i.e., type of contexts or type of objects) one image at each trial.
  Arms: semantic group
Other: Emotional group — The "emotional task" has to evaluate the emotional content (i.e., neutral, positive or negative) of one image at each trial.
  Arms: emotional group

SUMMARY:
The aim of this study is to analyse explicit and implicit emotional information processing abilities in children with attention deficit disorder with or without hyperactivity

DETAILED DESCRIPTION:
The main symptoms of Attentional Deficit Hyperactivity Disorder (ADHD) are inattention, motor agitation and impulsivity. However, other dysfunctions affecting the quality of life remain poorly studied: lack of understanding and management of emotions, focus on the local aspects of a visual scene limiting the ability to assign a general meaning to the scene and alteration of long-term memory encoding. This study aims to analyse these difficulties using different tasks requiring processing of rich and varied everyday images, having high ecological validity. It involves the participation of 56 boys and girls with ADHD, aged 7 to 12 years. A first phase examines the immediate understanding of images using two tasks: semantic categorization (Experiment 1) and emotional evaluation (Experiment 2) of images with positive, negative or neutral emotional valence, and depicting real environments (natural vs. manufactured contexts) or foreground objects pasted into a noise background (inanimate objects vs. animals vs. people. In each trial, one context image and one object image are presented briefly and simultaneously, one in each visual field. In order to be appropriately understood in both their semantic and emotional contents, context images will require more global processing, while object images will require more local, detailed processing. Their semantic (Exp. 1) and emotional (Exp. 2) consistency is manipulated. A week later, the participants have to perform a memory task requiring old/new recognition in a two-alternative forced choice (2AFC) paradigm that presents in each trial a pair of images (one old, one new) having the same emotional valence (Exp. 3). The study will characterize the specificities of processing and representing visual emotional information in ADHD children. The results will be compared with those from a previous study we conducted with the same methodology on neuro-typical children (controls).

ELIGIBILITY:
Inclusion Criteria:

* Children between 7 and 12 years old…………………………….
* Normal or corrected visual acuity ……………………………….
* ADHD diagnostic given by a doctor according to DSM 5 criteria (Diagnostic and Statistical Manual of Mental Disorders)
* Free from drug treatment until 24 hours before the experiment session……………………….
* Affiliation to a social security system…………………….
* Signature of the authorization documents from one parent or the holder of parental authority

Exclusion Criteria:

-History of neurological troubles, dysphasia, autistic spectrum disorder, intellectual disabilities

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2020-03-11 (Actual); Study Completion 2020-03-11 (Actual)

PRIMARY OUTCOMES:
1. Accuracy and response time at an explicit emotional evaluation task of visual scenes, by children with Attentional Deficit Hyperactivity Disorder (ADHD) | at baseline Day 0
  The performance at the emotional evaluation task is analyzed by association of two separate outcomes measures: measure of efficiency by the accuracy (i.e. proportion of correct response) and measure of the effectiveness by the response time at the correct trials (in milliseconds). This experiment analyzed the explicit processing of visual scenes' emotional content .
2. Accuracy and response time at a semantic categorization task of visual scenes, by children with Attentional Deficit Hyperactivity Disorder (ADHD) | at baseline Day 0
  The performance at the semantic categorization task is analyzed by association of two separate outcomes measures: measure of efficiency by the accuracy (i.e. proportion of correct response) and measure of the effectiveness by the response time at the correct trials (in milliseconds). This experiment analyzed the implicit processing of visual scenes' emotional content .

SECONDARY OUTCOMES:
Proportion and response time of correct response for the contextual images compared to the local images at the semantic categorization task for ADHD's participants | at baseline Day 0
  The performance is analyzed by association of two separate outcomes measures: measure of efficiency by the accuracy (i.e. proportion of correct response) and measure of the effectiveness by the response time at the correct trials (in milliseconds).
Proportion and response time of correct response for the contextual images compared to the local images at the emotional evaluation task for ADHD's participants | at baseline Day 0
  The performance is analyzed by association of two separate outcomes measures: measure of efficiency by the accuracy (i.e. proportion of correct response) and measure of the effectiveness by the response time at the correct trials (in milliseconds).
Influence of the image's emotional content (i.e. neutral, positive or negative) on long term memory in ADHD participants | at 1 week from the first evaluation
  The performance, in a two-alternative forced choice (2 AFC) image recognition, is analyzed by two separate outcomes measures: measure of efficiency by the accuracy (i.e. proportion of correct response) and measure of the effectiveness by the response time (in milliseconds).
Performance on long term memory in ADHD participants | at 1 week from the first evaluation
  The performance, in a two-alternative forced choice (2 AFC) image recognition, is analyzed by two separate outcomes measures: measure of efficiency by the accuracy (i.e. proportion of correct response) and measure of the effectiveness by the response time (in milliseconds).

CONTACTS AND LOCATIONS:
Overall Officials: FOSSOUD Catherine, MD, Principal Investigator — Fondation Lenval - Nice Children Hôpitaux Pédiatriques de Nice
Locations (1):
- Hôpitaux Pédiatriques de Nice CHU-Lenval, Nice, France